CLINICAL TRIAL: NCT01937975
Title: An Open-Label Study to Investigate the Pharmacokinetics of MK-5172 and MK-8742 in Subjects With Renal Insufficiency
Brief Title: The Pharmacokinetics of Grazoprevir (MK-5172) and Elbasvir (MK-8742) in Participants With Renal Insufficiency (MK-5172-050)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-050
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Chronic Hepatitis C; Renal Impairment
MeSH Terms: conditions — Hepatitis C, Chronic; Renal Insufficiency | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Participants with End Stage Renal Disease on Hemodialysis (Experimental): Participants with End Stage Renal Disease on hemodialysis received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days..
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Participants with Severe Renal Impairment (Experimental): Participants with Severe Renal Impairment (estimated glomerular filtration rate <30 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Healthy Participants (Experimental): Healthy participants (estimated glomerular filtration rate >=80 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir

INTERVENTIONS:
Drug: Grazoprevir — 100 mg oral tablet administered once a day for 10 days
Drug: Elbasvir — 50 mg oral tablet administered once a day for 10 days

SUMMARY:
Grazoprevir (MK-5172) and Elbasvir (MK-8742) were studied as the principal components of combination oral therapy for hepatitis C virus (HCV). The study examined the pharmacokinetic (PK) profiles of Grazoprevir and Elbasvir following 10 days of dosing in participants with end stage renal disease (ESRD) on hemodialysis (HD) or participants with severe renal impairment. Both groups were compared to healthy matched controls.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using an acceptable birth control method. Females of non-childbearing potential must have undergone a sterilization procedure at least 6 months prior to the first dose
* Non-vasectomized male participants must agree to use a condom with spermicide or abstain from sexual intercourse during the trial and for 90 days after stopping the study medication and agree not to donate sperm during this time period Participants with ESRD on HD
* Maintained on a stable regimen of HD within 3 months prior to first dosing Participants with Severe Renal Impairment
* Estimated glomerular filtration rate (eGFR) at screening is < 30 mL/min/1.73m^2 Healthy Controls
* Participant is within ± 10 years of the mean age and within 10% of the mean body mass index of severe renal impairment participants
* eGFR at screening is >=80 mL/min/1.73m^2

Exclusion Criteria:

All Participants

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease whose current condition is considered unstable
* History or presence of alcoholism and drug abuse within the past 6 months
* Female participants who are pregnant or lactating
* Regular user of any medication (including over the counter) that would significantly alter GFR
* Donation of blood or significant blood loss within 56 days prior to the first dose of study medication(s)
* Plasma donation within 7 days prior to the first dose of study medication(s)
* A renal transplant or nephrectomy Participants with ESRD or Severe Renal Impairment
* Rapidly fluctuating renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09-06 (Actual); Primary Completion 2013-12-17 (Actual); Study Completion 2013-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Caro L, Wenning L, Feng HP, Guo Z, Du L, Bhagunde P, Fandozzi C, Panebianco D, Marshall WL, Butterton JR, Iwamoto M, Yeh WW. Pharmacokinetics of elbasvir and grazoprevir in subjects with end-stage renal disease or severe renal impairment. Eur J Clin Pharmacol. 2019 May;75(5):665-675. doi: 10.1007/s00228-018-2585-3. Epub 2019 Jan 25. PMID 30680407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After enrollment of participants with End Stage Renal Disease and Severe Renal Impairment, healthy participants with matching mean age, body mass index, and gender were enrolled.
Period: Overall Study
Arm/Group | Participants With End Stage Renal Disease on Hemodialysis | Participants With Severe Renal Impairment | Healthy Participants
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With End Stage Renal Disease on Hemodialysis | Participants With Severe Renal Impairment | Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Full Range); unit: Years] | 47.8 [38 to 61] | 65.8 [54 to 75] | 55.1 [47 to 63] | 56.2 [38 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 5 | 4 | 4 | 13
Estimated Glomerular Filtration Rate [Mean (Full Range); unit: mL/min/1.73 m^2] — Glomerular Filtration Rate at baseline was based on the Modification of Diet Renal Disease equation. N=6 instead of 8 for Healthy Participants.
  mL/min/1.73 m^2 | NA [NA to NA] — Not determined for ESRD participants on HD | 18.0 [11.5 to 23.5] | 93.4 [80.0 to 124.0] | NA [NA to NA] — Not determined for the overall population

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours Postdose (AUC0-24hr) of Grazoprevir
Description: Blood for determination of Grazoprevir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, and 24 hours postdose on Day 9 (ESRD participants only) or Day 10 (all participants)
Time Frame: Up to 24 hours postdose
Population: The Per Protocol population included all participants who complied with the protocol sufficiently to ensure that these data likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Groups:
- Participants With End Stage Renal Disease: Participants with End Stage Renal Disease (ESRD) on hemodialysis (HD) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days. Day 9 was a non-hemodialysis day for these participants. On Day 10, hemodialysis for these participants was timed to occur after the median Tmax (~5 hours postdose).
- Participants With Severe Renal Impairment: Day 10: Participants with Severe Renal Impairment (SRI, estimated glomerular filtration rate <30 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days.
- Healthy Participants: Day 10: Healthy participants (estimated glomerular filtration rate >=80 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days.
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
uM*hr
  Day 9 | 0.969 [0.689 to 1.36] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 0.944 [0.671 to 1.33] | 1.88 [1.23 to 2.86] | 1.14 [0.843 to 1.54]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.97, 90% CI 2-sided [0.87 to 1.09] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.85, 90% CI 2-sided [0.58 to 1.25] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.83, 90% CI 2-sided [0.56 to 1.22] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.65, 90% CI 2-sided [1.09 to 2.49] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

2. Primary Outcome: Plasma Concentration at 24 Hours Postdose (C24hr) of Grazoprevir
Description: Blood for determination of Grazoprevir concentration was collected at 24 hours postdose on Day 9 (ESRD participants only) or Day 10 (all participants)
Time Frame: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Groups:
- Participants With Severe Renal Impairment: Day 10: Participants with Severe Renal Impairment (estimated glomerular filtration rate <30 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days.
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
nM
  Day 9 | 11.4 [8.16 to 16.1] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 11.3 [8.03 to 15.8] | 23.3 [15.4 to 35.2] | 14.5 [10.7 to 19.6]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.81 to 1.19] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.79, 90% CI 2-sided [0.54 to 1.16] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.78, 90% CI 2-sided [0.53 to 1.14] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.60, 90% CI 2-sided [1.06 to 2.42] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Grazoprevir
Description: Blood for determination of Grazoprevir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, 24, 32, 48, 72, 96, and 120 hours postdose on Day 10 (all participants) and only up to 24 hours for ESRD participants on Day 9
Time Frame: Up to 120 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: uM
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
uM
  Day 9 | 0.141 [0.092 to 0.215] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 0.135 [0.088 to 0.206] | 0.255 [0.152 to 0.429] | 0.154 [0.106 to 0.224]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.96, 90% CI 2-sided [0.75 to 1.22] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.57 to 1.48] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.88, 90% CI 2-sided [0.54 to 1.42] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.66, 90% CI 2-sided [0.99 to 2.77] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

4. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Grazoprevir
Description: as for outcome 3
Time Frame: Up to 120 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Hours
  Day 9 | 2.00 [1.00 to 6.00] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 2.50 [0.50 to 7.00] | 3.00 [0.50 to 6.00] | 2.50 [1.00 to 6.00]

5. Primary Outcome: Apparent Terminal Half-life (T1/2) of Grazoprevir
Description: Blood for determination of Grazoprevir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, 24, 32, 48, 72, 96, and 120 hours postdose on Day 10
Time Frame: Up to 120 hours postdose
Population: The Per Protocol population included all participants who complied with the protocol sufficiently to ensure that these data likely to exhibit the effects of treatment, according to the underlying scientific model. End Stage Renal Disease for Non-HD Day 9 was not reported since only 24-hour collections were made on that day.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Groups:
- Participants With End Stage Renal Disease: HD Day 10: Participants with End Stage Renal Disease (ESRD) on hemodialysis (HD) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days. Day 9 was a non-hemodialysis day for these participants. On Day 10, hemodialysis for these participants was timed to occur after the median Tmax (~5 hours postdose).
Arm/Group | Participants With End Stage Renal Disease: HD Day 10 | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Hours | 28.38 (20.88) [0.50 to 6.00] | 36.30 (30.53) [1.00 to 6.00] | 35.18 (19.64)

6. Primary Outcome: Apparent Clearance After Extravascular Administration (CL/F) of Grazoprevir
Description: as for outcome 1
Time Frame: Up to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/hr
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Liters/hr
  Day 9 | 135 [95.6 to 189] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 138 [98.1 to 194] | 69.4 [45.6 to 106] | 114 [84.5 to 155]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.92 to 1.15] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.18, 90% CI 2-sided [0.80 to 1.73] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.21, 90% CI 2-sided [0.82 to 1.78] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.61, 90% CI 2-sided [0.40 to 0.92] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

7. Primary Outcome: Apparent Volume of Distribution After Extravascular Administration (Vz/F) of Grazoprevir
Description: Blood for determination of Grazoprevir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, and 24 hours postdose on Day 10
Time Frame: Up to 24 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Participants With End Stage Renal Disease: HD Day 10 | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Liters | 5430 [3660 to 8050] | 3490 [2320 to 5260] | 5760 [4180 to 7930]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease: HD Day 10 vs Healthy Participants: Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.63 to 1.42] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 2: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.61, 90% CI 2-sided [0.39 to 0.94] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

8. Primary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours Postdose (AUC0-24hr) of Elbasvir
Description: Blood for determination of Elbasvir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, and 24 hours postdose on Day 9 (ESRD participants only) or Day 10 (all participants)
Time Frame: Up to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: uM*hr
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
uM*hr
  Day 9 | 1.89 [1.48 to 2.42] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 2.16 [1.69 to 2.77] | 4.07 [3.01 to 5.52] | 2.19 [1.76 to 2.72]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.14, 90% CI 2-sided [1.08 to 1.21] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.86, 90% CI 2-sided [0.65 to 1.14] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.75 to 1.30] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.86, 90% CI 2-sided [1.38 to 2.51] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

9. Primary Outcome: Plasma Concentration at 24 Hours Postdose (C24hr) of Elbasvir
Description: Blood for determination of Elbasvir concentration was collected at 24 hours postdose on Day 9 (ESRD participants only) or Day 10 (all participants)
Time Frame: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
nM
  Day 9 | 46.9 [35.2 to 62.4] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 58.2 [43.7 to 77.5] | 126 [88.6 to 179] | 60.9 [47.3 to 78.5]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.24, 90% CI 2-sided [1.17 to 1.32] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.77, 90% CI 2-sided [0.56 to 1.06] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.95, 90% CI 2-sided [0.69 to 1.32] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 2.07, 90% CI 2-sided [1.46 to 2.93] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

10. Primary Outcome: Maximum Plasma Concentration (Cmax) of Elbasvir
Description: Blood for determination of Elbasvir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, 24, 32, 48, 72, 96, and 120 hours postdose on Day 10 (all participants) and only up to 24 hours for ESRD participants on Day 9
Time Frame: Up to 120 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: uM
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
uM
  Day 9 | 0.137 [0.105 to 0.178] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 0.154 [0.118 to 0.200] | 0.271 [0.196 to 0.373] | 0.163 [0.129 to 0.206]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.12, 90% CI 2-sided [1.00 to 1.26] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.84, 90% CI 2-sided [0.62 to 1.13] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.70 to 1.27] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.66, 90% CI 2-sided [1.21 to 2.28] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

11. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Elbasvir
Description: as for outcome 10
Time Frame: Up to 120 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Hours
  Day 9 | 4.00 [3.00 to 4.00] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 5.00 [3.00 to 5.00] | 4.00 [4.00 to 6.00] | 4.00 [2.00 to 4.00]

12. Primary Outcome: Apparent Terminal Half-life (T1/2) of Elbasvir
Description: Blood for determination of Elbasvir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, 24, 32, 48, 72, 96, and 120 hours postdose on Day 10
Time Frame: Up to 120 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Groups:
- Healthy Participants: Day 10: Healthy participants (estimated glomerular filtration rate >=80 mL/min/1.73 m^2) received once daily Grazoprevir 100 mg tablet and Elbasvir 50 mg tablet for 10 days. One participant was excluded due to an ill-defined terminal phase.
Arm/Group | Participants With End Stage Renal Disease: HD Day 10 | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 7
Hours | 23.04 (6.34) [0.50 to 6.00] | 28.97 (18.26) [1.00 to 6.00] | 25.02 (19.08)

13. Primary Outcome: Apparent Clearance After Extravascular Administration (CL/F) of Elbasvir
Description: as for outcome 8
Time Frame: Up to 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/hr
Arm/Group | Participants With End Stage Renal Disease | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 8
Liters/hr
  Day 9 | 29.9 [23.4 to 38.3] | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group | NA [NA to NA] — No pharmacokinetic sampling on Day 9 for this group
  Day 10 | 26.2 [20.5 to 33.5] | 13.9 [10.3 to 18.9] | 25.9 [20.8 to 32.2]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease; ESRD Non-HD Day 9 versus ESRD HD Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.88, 90% CI 2-sided [0.83 to 0.92] — Geometric Mean Ratio = ESRD HD Day 10 / ESRD Non-HD Day 9
Statistical Analysis 2: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD Non-HD Day 9 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.16, 90% CI 2-sided [0.88 to 1.53] — Geometric Mean Ratio = ESRD Non-HD Day 9 / Healthy Day 10
Statistical Analysis 3: Comparison: Participants With End Stage Renal Disease vs Healthy Participants: Day 10; ESRD HD Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 1.01, 90% CI 2-sided [0.77 to 1.34] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 4: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; SRI Participants Day 10 versus Healthy Participants Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.54, 90% CI 2-sided [0.40 to 0.72] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

14. Primary Outcome: Apparent Volume of Distribution After Extravascular Administration (Vz/F) of Elbasvir
Description: Blood for determination of Elbasvir concentration was collected predose and 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 12, 16, and 24 hours postdose on Day 10
Time Frame: Up to 24 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Participants With End Stage Renal Disease: HD Day 10 | Participants With Severe Renal Impairment: Day 10 | Healthy Participants: Day 10
Number analyzed (Participants) | 8 | 8 | 7
Liters | 857 [641 to 1150] | 569 [420 to 772] | 901 [699 to 1160]
Statistical Analysis 1: Comparison: Participants With End Stage Renal Disease: HD Day 10 vs Healthy Participants: Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.95, 90% CI 2-sided [0.70 to 1.30] — Geometric Mean Ratio = ESRD HD Day 10 / Healthy Day 10
Statistical Analysis 2: Comparison: Participants With Severe Renal Impairment: Day 10 vs Healthy Participants: Day 10; Test type: Superiority or Other; Geometric Mean Ratio = 0.63, 90% CI 2-sided [0.45 to 0.89] — Geometric Mean Ratio = SRI Day 10 / Healthy Day 10

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (up to 24 days)
Arm/Group | Participants With End Stage Renal Disease on Hemodialysis | Participants With Severe Renal Impairment | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With End Stage Renal Disease on Hemodialysis (N=8) | Participants With Severe Renal Impairment (N=8) | Healthy Participants (N=8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will provide separate guidance on the criteria for publication of clinical trial data when contacted for permission to publish.